CLINICAL TRIAL: NCT02980731
Title: Open-Label, Single Arm, Phase 3b, Multi-Center Study Evaluating the Impact of Venetoclax on the Quality of Life of Relapsed/Refractory Subjects With Chronic Lymphocytic Leukemia (CLL) (VENICE II)
Brief Title: A Study Evaluating the Impact of Venetoclax on the Quality of Life for Subjects With Relapsed (Your Cancer Has Come Back) or Refractory (no Response to Previous Cancer Treatments) Chronic Lymphocytic Leukemia (CLL) While Receiving Venetoclax Monotherapy (a Single Agent).
Acronym: VENICE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-889; 2016-001097-15 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Relapsed CLL; Refractory CLL; 17p deletion; TP53 gene; B-Cell receptor inhibitor (BCRi); European Organization of Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30); Overall response rate (ORR); Duration of overall response (DOR); Complete remission rate (CR + CRi); Progression-free survival (PFS); Overall survival (OS)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Venetoclax (Experimental): Venetoclax was administered orally once daily (QD) for a planned duration of up to 2 years or until disease progression; median time on treatment was 127 weeks. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Venetoclax tablets were to be taken orally once daily with a meal and water in the morning at approximately the same time each day. Tablets were to be swallowed whole and not chewed, crushed, or broken prior to swallowing.
  Other Names: ABT-199; VENCLEXTA; VENCLYXTO

SUMMARY:
The purpose of this open-label, single-arm study was to evaluate the impact of venetoclax on the quality of life of participants including those with with relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL; a type of cancer affecting the blood and the bone marrow) with or without the 17p deletion or TP53 mutation, including participants with an unknown status, as well as R/R CLL participants who had been previously treated with B-cell receptor inhibitor (BCRi) therapy. The starting dose of venetoclax was 20 mg once daily. The dose must have been gradually increased over a period of 5 weeks up to the daily dose of 400 mg. Participants may have continued receiving venetoclax for up to 2 years. After the treatment period, participants may have continued on into a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2
* Participant has relapsed/refractory disease (received at least one prior therapy)
* Diagnosis of CLL that meets published 2008 Modified International Workshop on CLL National Cancer Institute - Working Group (IWCLL NCI-WG) Guidelines and:

  * has an indication for treatment according to the 2008 Modified IWCLL NCI-WG Guidelines
  * has clinically measurable disease (lymphocytosis > 5 × 10^9/L and/or palpable and measurable nodes by physical exam and/or organomegaly assessed by physical exam)
  * with or without 17p deletion or TP53 mutation
  * may have been previously treated with a prior B-cell receptor inhibitor therapy
* Adequate bone marrow function

Exclusion Criteria:

* Participant has developed Richter's transformation or Prolymphocytic leukemia (PLL)
* Participant has previously received venetoclax
* History of active malignancies other than CLL within the past 2 years prior to first dose of venetoclax, with the exception of:

  * adequately treated in situ carcinoma of the cervix uteri
  * adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
  * previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
* Active and uncontrolled autoimmune cytopenias (within 2 weeks prior to screening), including autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP), despite low dose corticosteroids
* Prior allogeneic stem cell transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (33):
- Argentina (4):
  - Hospital Italiano La Plata /ID# 150812, La Plata, Buenos Aires
  - Fundaleu /Id# 150811, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Cemic /Id# 150810, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Sanatorio Allende /ID# 150813, Córdoba
- Australia (5):
  - St George Hospital /ID# 154212, Kogarah, New South Wales
  - Liverpool Hospital /ID# 154950, Liverpool, New South Wales
  - Gold coast University Hospital /ID# 150833, Southport, Queensland
  - Peter MacCallum Cancer Ctr /ID# 154948, Melbourne, Victoria
  - Perth Blood Institute Ltd /ID# 154949, Nedlands, Western Australia
- Bulgaria (4):
  - UMHAT Alexandrovska EAD /ID# 162987, Sofiya, Sofia
  - UMHAT Sveti Georgi /ID# 161594, Plovdiv
  - UMHAT Sveti Ivan Rilski /ID# 163280, Sofia
  - SHAT Hematologic Diseases /ID# 161592, Sofia
- Hong Kong (2):
  - Prince of Wales Hospital /ID# 150837, Hong Kong
  - Queen Mary Hospital /ID# 150836, Hong Kong
- Hungary (2):
  - Semmelweis Egyetem /ID# 150792, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 152842, Budapest
- Mexico (2):
  - Centro de Investigacion Clínica Chapultepec SA de CV /ID# 163641, Morelia, Michoacán
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 150821, Monterrey, Nuevo León
- New Zealand (3):
  - Middlemore Clinical Trials /ID# 161526, Papatoetoe, Auckland
  - North Shore Hospital /ID# 157626, Takapuna, Auckland
  - Wellington Regional Hospital /ID# 157627, Newtown, Wellington Region
- Poland (4):
  - Instytut Hematologii i Transfuzjologii /ID# 150878, Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o.o /ID# 164097, Gdynia, Pomeranian Voivodeship
  - SP ZOZ Zespol Szpitali Miejskich w Chorzowie /ID# 150877, Chorzów, Silesian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopern /ID# 150880, Lodz, Łódź Voivodeship
- Russia (4):
  - Federal State Budgetary Scientific Institution N.N. Blokhin /ID# 166610, Moscow, Moscow
  - Moscow State budget healthcare /ID# 154806, Moscow, Moscow
  - Regional Oncological Dispensary /ID# 154202, Penza, Penza Oblast
  - Federal State Budgetary Ins NRC for Hematology of MoH of Russian Federation /ID# 154213, Moscow
- Taiwan (3):
  - China Medical University Hospital /ID# 150839, Taichung
  - National Taiwan University Hospital /ID# 150838, Taipei
  - Taipei Veterans General Hosp /ID# 153803, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Cochrane T, Enrico A, Gomez-Almaguer D, Hadjiev E, Lech-Maranda E, Masszi T, Nikitin E, Robak T, Weinkove R, Wu SJ, Sail KR, Pesko J, Pai M, Komlosi V, Anderson MA. Impact of venetoclax monotherapy on the quality of life of patients with relapsed or refractory chronic lymphocytic leukemia: results from the phase 3b VENICE II trial. Leuk Lymphoma. 2022 Feb;63(2):304-314. doi: 10.1080/10428194.2021.1986217. Epub 2021 Oct 11. PMID 34632935

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants who received at least one dose of venetoclax
Period: Overall Study
Arm/Group | Venetoclax
Started | 210
Completed | 0
Not Completed | 210
Not completed — Death | 63
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 5
Not completed — Study terminated by Sponsor | 4
Not completed — Completed survival follow-up period | 65
Not completed — COVID-19 infection | 1
Not completed — Other, not specified | 66

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of venetoclax
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 141
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 182
  Black or African American | 1
  Asian | 18
  American Indian or Alaska Native | 8
  Native Hawaiian or other Pacific Islander | 1
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 48 in Global Health Status/Quality of Life (GHS/QoL) Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the global health status/quality of life scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: Baseline, Week 48
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 157
units on a scale | 9.3 (20.11)
Statistical Analysis 1: Comparison: Venetoclax; Test type: Superiority; p = 0.004, t-test, 2 sided — P-value is derived from a paired t-test of H0: mean difference (Week 48 - baseline) ≤ 5 versus H1: mean difference (Week 48 - baseline) > 5

2. Secondary Outcome: Mean Change From Baseline in Global Health Status/Quality of Life (GHS/QoL) Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, Final visit (at study drug discontinuation and/or upon discontinuation from the study, up to Week 108)
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | 3.9 (17.65)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 6.0 (20.67)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 7.6 (20.13)
  Week 24: number analyzed (Participants) | 179
  Week 24 | 9.2 (20.29)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 9.4 (19.45)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 9.3 (20.11)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 10.3 (21.83)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 10.2 (23.87)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 11.2 (20.96)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 8.9 (20.92)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 9.2 (19.97)
  Final visit | 4.8 (23.58)

3. Secondary Outcome: Mean Change From Baseline in Physical Functioning Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a physical functioning scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the physical functioning scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | 1.2 (12.86)
  Week 8: number analyzed (Participants) | 189
  Week 8 | 3.0 (16.16)
  Week 12: number analyzed (Participants) | 190
  Week 12 | 4.6 (15.89)
  Week 24: number analyzed (Participants) | 181
  Week 24 | 5.2 (16.90)
  Week 36: number analyzed (Participants) | 168
  Week 36 | 5.6 (15.59)
  Week 48: number analyzed (Participants) | 158
  Week 48 | 6.1 (16.30)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 6.0 (17.73)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 5.7 (18.47)
  Week 84: number analyzed (Participants) | 140
  Week 84 | 4.8 (15.04)
  Week 96: number analyzed (Participants) | 135
  Week 96 | 4.0 (17.18)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 5.7 (16.43)
  Final visit | 1.8 (20.52)

4. Secondary Outcome: Mean Change From Baseline in Role Functioning Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a role functioning scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the role functioning scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | 2.6 (22.75)
  Week 8: number analyzed (Participants) | 189
  Week 8 | 4.0 (28.31)
  Week 12: number analyzed (Participants) | 190
  Week 12 | 7.1 (28.60)
  Week 24: number analyzed (Participants) | 180
  Week 24 | 9.2 (26.85)
  Week 36: number analyzed (Participants) | 168
  Week 36 | 9.8 (26.70)
  Week 48: number analyzed (Participants) | 158
  Week 48 | 10.4 (26.10)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 8.4 (27.63)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 11.6 (31.01)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 9.9 (27.38)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 8.3 (31.23)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 11.5 (28.03)
  Final visit | 3.3 (33.29)

5. Secondary Outcome: Mean Change From Baseline in Emotional Functioning Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including an emotional functioning scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the emotional functioning scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | 4.9 (16.30)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 4.7 (16.96)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 5.7 (17.11)
  Week 24: number analyzed (Participants) | 179
  Week 24 | 3.6 (17.62)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 4.3 (17.08)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 5.7 (17.64)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 5.2 (18.79)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 5.1 (18.54)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 4.0 (17.95)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 4.2 (19.95)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 6.1 (20.18)
  Final visit | 1.4 (21.78)

6. Secondary Outcome: Mean Change From Baseline in Cognitive Functioning Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a cognitive functioning scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the cognitive functioning scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | 2.3 (15.61)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 4.2 (18.93)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 4.3 (18.29)
  Week 24: number analyzed (Participants) | 179
  Week 24 | 3.4 (18.42)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 3.8 (18.54)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 3.7 (17.15)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 4.1 (20.01)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 4.7 (17.65)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 3.5 (17.91)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 1.1 (19.58)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 5.6 (18.75)
  Final visit | 2.3 (20.79)

7. Secondary Outcome: Mean Change From Baseline in Social Functioning Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a social functioning scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the social functioning scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | 2.2 (19.14)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 5.5 (22.13)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 6.6 (22.26)
  Week 24: number analyzed (Participants) | 179
  Week 24 | 7.2 (24.79)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 8.6 (21.63)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 9.9 (22.80)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 9.2 (25.78)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 9.7 (27.41)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 8.7 (23.95)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 8.2 (26.14)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 11.7 (24.21)
  Final visit | 3.4 (29.70)

8. Secondary Outcome: Mean Change From Baseline in Fatigue Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a fatigue scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the fatigue scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -4.6 (18.63)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -7.7 (22.70)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -11.2 (24.66)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -10.9 (20.70)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -12.5 (23.21)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -12.9 (21.40)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -13.0 (22.79)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -13.8 (25.90)
  Week 84: number analyzed (Participants) | 140
  Week 84 | -12.9 (23.49)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -10.7 (24.13)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -13.8 (22.69)
  Final visit | -7.5 (26.16)

9. Secondary Outcome: Mean Change From Baseline in Nausea and Vomiting Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a nausea and vomiting scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the nausea and vomiting scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -0.2 (18.02)
  Week 8: number analyzed (Participants) | 189
  Week 8 | 0.4 (17.19)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -0.3 (18.50)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -1.5 (17.24)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -2.0 (16.19)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -0.6 (19.45)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -0.3 (15.42)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 0.3 (17.40)
  Week 84: number analyzed (Participants) | 139
  Week 84 | 0.4 (18.00)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 0.1 (17.15)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -1.1 (16.28)
  Final visit | -0.8 (17.58)

10. Secondary Outcome: Mean Change From Baseline in Pain Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a pain scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the pain scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -4.6 (21.05)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -2.9 (21.31)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -3.6 (22.56)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -4.1 (22.08)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -4.0 (22.43)
  Week 48: number analyzed (Participants) | 157
  Week 48 | -4.6 (20.29)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -5.2 (23.46)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -4.7 (23.30)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -4.6 (22.10)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 1.1 (25.35)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -3.4 (24.33)
  Final visit | -0.1 (26.50)

11. Secondary Outcome: Mean Change From Baseline in Dyspnea Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a dyspnea scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the dyspnea scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -3.7 (23.33)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -5.5 (26.62)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -7.7 (29.08)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -8.5 (26.56)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -8.3 (28.43)
  Week 48: number analyzed (Participants) | 157
  Week 48 | -8.5 (27.19)
  Week 60: number analyzed (Participants) | 153
  Week 60 | -8.5 (26.08)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -9.2 (31.30)
  Week 84: number analyzed (Participants) | 140
  Week 84 | -9.3 (26.84)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -6.4 (28.55)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -10.9 (27.92)
  Final visit | -5.3 (29.60)

12. Secondary Outcome: Mean Change From Baseline in Insomnia Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including an insomnia scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the insomnia scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -6.5 (25.78)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -7.9 (30.39)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -9.1 (29.27)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -9.0 (27.19)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -8.3 (30.68)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -11.6 (25.77)
  Week 60: number analyzed (Participants) | 153
  Week 60 | -10.2 (28.94)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -7.8 (29.40)
  Week 84: number analyzed (Participants) | 140
  Week 84 | -9.5 (28.35)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -6.6 (29.76)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -10.7 (26.16)
  Final visit | -5.3 (30.52)

13. Secondary Outcome: Mean Change From Baseline in Appetite Loss Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including an appetite loss scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the appetite loss scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -3.4 (23.63)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -6.2 (24.85)
  Week 12: number analyzed (Participants) | 189
  Week 12 | -6.0 (29.56)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -8.8 (27.36)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -8.1 (24.06)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -7.8 (24.14)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -5.6 (27.16)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -5.1 (27.59)
  Week 84: number analyzed (Participants) | 140
  Week 84 | -6.9 (24.16)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -6.4 (27.07)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -9.3 (25.81)
  Final visit | -4.0 (30.36)

14. Secondary Outcome: Mean Change From Baseline in Constipation Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a constipation scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the constipation scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | 1.7 (17.87)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 2.5 (21.38)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 1.4 (20.58)
  Week 24: number analyzed (Participants) | 180
  Week 24 | 1.1 (18.61)
  Week 36: number analyzed (Participants) | 167
  Week 36 | -0.8 (20.36)
  Week 48: number analyzed (Participants) | 156
  Week 48 | -0.2 (18.35)
  Week 60: number analyzed (Participants) | 153
  Week 60 | 1.7 (20.52)
  Week 72: number analyzed (Participants) | 143
  Week 72 | 0.5 (18.97)
  Week 84: number analyzed (Participants) | 138
  Week 84 | 1.7 (19.45)
  Week 96: number analyzed (Participants) | 135
  Week 96 | 0.7 (20.55)
  Week 108: number analyzed (Participants) | 121
  Week 108 | -0.8 (18.98)
  Final visit | 1.2 (19.64)

15. Secondary Outcome: Mean Change From Baseline in Diarrhea Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a diarrhea scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the diarrhea scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | -0.7 (20.63)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 1.8 (21.45)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 2.3 (22.30)
  Week 24: number analyzed (Participants) | 179
  Week 24 | 4.7 (21.42)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 4.6 (21.62)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 4.0 (21.13)
  Week 60: number analyzed (Participants) | 154
  Week 60 | 7.4 (27.01)
  Week 72: number analyzed (Participants) | 145
  Week 72 | 3.0 (25.74)
  Week 84: number analyzed (Participants) | 141
  Week 84 | 4.3 (23.18)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 3.7 (22.47)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 3.8 (21.51)
  Final visit | 4.9 (23.30)

16. Secondary Outcome: Mean Change From Baseline in Financial Difficulties Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item participant self-report questionnaire composed of both multi-item and single scales, including a financial difficulties scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the financial difficulties scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | -6.4 (20.07)
  Week 8: number analyzed (Participants) | 187
  Week 8 | -4.6 (21.91)
  Week 12: number analyzed (Participants) | 189
  Week 12 | -6.0 (24.54)
  Week 24: number analyzed (Participants) | 179
  Week 24 | -7.3 (25.05)
  Week 36: number analyzed (Participants) | 167
  Week 36 | -7.8 (23.70)
  Week 48: number analyzed (Participants) | 157
  Week 48 | -8.9 (26.52)
  Week 60: number analyzed (Participants) | 153
  Week 60 | -10.0 (25.96)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -8.5 (27.99)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -10.9 (23.06)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -8.6 (25.34)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -9.6 (24.04)
  Final visit | -6.5 (25.88)

17. Secondary Outcome: Mean Change From Baseline in Fatigue Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the fatigue scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -6.3 (32.20)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -10.2 (38.11)
  Week 12: number analyzed (Participants) | 189
  Week 12 | -13.9 (38.59)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -15.3 (37.96)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -16.3 (34.41)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -16.1 (35.41)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -14.5 (36.59)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -16.4 (36.85)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -17.4 (34.90)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -13.0 (35.18)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -19.8 (35.17)
  Final visit | -10.6 (41.71)

18. Secondary Outcome: Mean Change From Baseline in Treatment Side Effects Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the treatment side effects scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -2.6 (17.70)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -4.0 (17.84)
  Week 12: number analyzed (Participants) | 189
  Week 12 | -4.8 (17.96)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -7.5 (18.46)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -7.8 (18.03)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -7.5 (19.19)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -6.3 (19.41)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -6.3 (18.73)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -6.8 (16.43)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -6.9 (18.48)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -8.2 (19.33)
  Final visit | -3.6 (22.54)

19. Secondary Outcome: Mean Change From Baseline in Disease Effects Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the disease effects scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -10.7 (19.58)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -10.0 (21.80)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -12.4 (23.48)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -13.7 (23.63)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -13.9 (23.34)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -13.4 (23.68)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -13.1 (23.18)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -13.8 (23.22)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -13.6 (22.69)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -13.2 (22.59)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -15.6 (24.93)
  Final visit | -10.2 (25.97)

20. Secondary Outcome: Mean Change From Baseline in Infection Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the infection scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 200
units on a scale
  Week 4: number analyzed (Participants) | 196
  Week 4 | -3.5 (21.66)
  Week 8: number analyzed (Participants) | 189
  Week 8 | -6.0 (29.00)
  Week 12: number analyzed (Participants) | 190
  Week 12 | -4.6 (28.67)
  Week 24: number analyzed (Participants) | 181
  Week 24 | -6.1 (26.50)
  Week 36: number analyzed (Participants) | 168
  Week 36 | -8.9 (26.04)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -9.0 (25.54)
  Week 60: number analyzed (Participants) | 154
  Week 60 | -7.9 (25.13)
  Week 72: number analyzed (Participants) | 145
  Week 72 | -8.5 (28.97)
  Week 84: number analyzed (Participants) | 141
  Week 84 | -9.9 (24.18)
  Week 96: number analyzed (Participants) | 136
  Week 96 | -8.5 (25.34)
  Week 108: number analyzed (Participants) | 122
  Week 108 | -10.3 (25.41)
  Final visit | -5.5 (29.97)

21. Secondary Outcome: Mean Change From Baseline in Social Problems Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the social problems scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 198
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | -4.0 (37.50)
  Week 8: number analyzed (Participants) | 187
  Week 8 | -7.5 (39.15)
  Week 12: number analyzed (Participants) | 188
  Week 12 | -8.5 (41.06)
  Week 24: number analyzed (Participants) | 179
  Week 24 | -10.6 (41.72)
  Week 36: number analyzed (Participants) | 166
  Week 36 | -13.7 (38.15)
  Week 48: number analyzed (Participants) | 156
  Week 48 | -15.6 (40.85)
  Week 60: number analyzed (Participants) | 152
  Week 60 | -15.6 (37.18)
  Week 72: number analyzed (Participants) | 143
  Week 72 | -17.5 (42.76)
  Week 84: number analyzed (Participants) | 139
  Week 84 | -15.3 (42.14)
  Week 96: number analyzed (Participants) | 134
  Week 96 | -14.7 (41.79)
  Week 108: number analyzed (Participants) | 120
  Week 108 | -16.1 (43.85)
  Final visit | -4.0 (48.50)

22. Secondary Outcome: Mean Change From Baseline in Future Health Subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chronic Lymphocytic Leukemia Module (EORTC QLQ-CLL16)
Description: EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life important in CLL. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the future health scale indicates a lower level of functioning, and negative changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 198
units on a scale
  Week 4: number analyzed (Participants) | 194
  Week 4 | -17.2 (37.82)
  Week 8: number analyzed (Participants) | 187
  Week 8 | -21.6 (42.94)
  Week 12: number analyzed (Participants) | 188
  Week 12 | -25.5 (41.77)
  Week 24: number analyzed (Participants) | 180
  Week 24 | -23.0 (38.96)
  Week 36: number analyzed (Participants) | 167
  Week 36 | -24.4 (43.97)
  Week 48: number analyzed (Participants) | 156
  Week 48 | -24.1 (41.75)
  Week 60: number analyzed (Participants) | 153
  Week 60 | -25.1 (46.09)
  Week 72: number analyzed (Participants) | 144
  Week 72 | -27.8 (40.59)
  Week 84: number analyzed (Participants) | 140
  Week 84 | -20.7 (39.68)
  Week 96: number analyzed (Participants) | 135
  Week 96 | -24.9 (44.18)
  Week 108: number analyzed (Participants) | 121
  Week 108 | -23.7 (46.63)
  Final visit | -16.7 (49.90)

23. Secondary Outcome: Mean Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale Score
Description: The EQ-5D 5L measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on five levels of severity (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems), and a separate visual analog scale (VAS). Participants rated their health on a vertical visual analogue scale, where the endpoints were labelled 100, "The best health you can imagine" and 0, "The worst health you can imagine". Positive values indicate improvement from baseline.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 199
units on a scale
  Week 4: number analyzed (Participants) | 195
  Week 4 | 3.67 (12.683)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 6.00 (15.982)
  Week 12: number analyzed (Participants) | 189
  Week 12 | 7.75 (14.498)
  Week 24: number analyzed (Participants) | 181
  Week 24 | 7.78 (16.158)
  Week 36: number analyzed (Participants) | 167
  Week 36 | 9.08 (16.342)
  Week 48: number analyzed (Participants) | 157
  Week 48 | 10.34 (16.808)
  Week 60: number analyzed (Participants) | 153
  Week 60 | 10.84 (17.180)
  Week 72: number analyzed (Participants) | 144
  Week 72 | 11.19 (17.890)
  Week 84: number analyzed (Participants) | 140
  Week 84 | 10.22 (15.431)
  Week 96: number analyzed (Participants) | 134
  Week 96 | 9.98 (16.310)
  Week 108: number analyzed (Participants) | 120
  Week 108 | 10.77 (17.500)
  Final Visit | 6.22 (19.262)

24. Secondary Outcome: Mean Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Health Index Score
Description: The EQ-5D 5L measures quality of life in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on five levels of severity (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems), and a separate visual analog scale (VAS). The scores for the 5 dimensions are used to compute a single utility index score ranging from zero (0.0) to 1 (1.0) representing the general health status of the individual, with '0' defined as a health state equivalent to being dead and '1' is full health. The higher the score the better the health status. Positive values indicate improvement from baseline.
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of venetoclax with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 201
units on a scale
  Week 4: number analyzed (Participants) | 197
  Week 4 | 0.02 (0.135)
  Week 8: number analyzed (Participants) | 190
  Week 8 | 0.02 (0.130)
  Week 12: number analyzed (Participants) | 191
  Week 12 | 0.03 (0.122)
  Week 24: number analyzed (Participants) | 183
  Week 24 | 0.03 (0.112)
  Week 36: number analyzed (Participants) | 168
  Week 36 | 0.04 (0.121)
  Week 48: number analyzed (Participants) | 159
  Week 48 | 0.04 (0.124)
  Week 60: number analyzed (Participants) | 155
  Week 60 | 0.04 (0.129)
  Week 72: number analyzed (Participants) | 146
  Week 72 | 0.03 (0.132)
  Week 84: number analyzed (Participants) | 142
  Week 84 | 0.03 (0.111)
  Week 96: number analyzed (Participants) | 136
  Week 96 | 0.01 (0.134)
  Week 108: number analyzed (Participants) | 122
  Week 108 | 0.02 (0.124)
  Final Visit | -0.01 (0.172)

25. Secondary Outcome: Complete Remission Rate (Complete Remission [CR] + Complete Remission With Incomplete Marrow Recovery [CRi])
Description: Complete remission rate (CR + CRi) is defined as the percentage of participants achieving a CR or CRi as their best response (per the investigator assessment) based on 2008 Modified International Workshop on Chronic Lymphocytic Leukemia (IWCLL) National Cancer Institute-Working Group (NCI-WG) Guidelines criteria.
Time Frame: From the first dose of study drug until the last participant completed the Week 48 assessments; median time on follow-up was 184 weeks
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
percentage of participants | 18.6 [13.6 to 24.5]

26. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved complete remission (CR), complete remission with incomplete marrow recovery (CRi), nodular partial remission (nPR), or confirmed partial remission (PR) based on the 2008 Modified International Workshop on Chronic Lymphocytic Leukemia (IWCLL) National Cancer Institute-Working Group (NCI-WG) Guidelines criteria as assessed by investigator using the best response at any time during the study.
Time Frame: as for outcome 25
Population: All enrolled participants who received at least one dose of venetoclax; participants who did not respond were considered non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
percentage of participants | 76.7 [70.4 to 82.2]

27. Secondary Outcome: Duration of Overall Response (DOR)
Description: DoR is defined as the number of days from the date of first response (complete remission (CR), complete remission with incomplete marrow recovery (CRi), nodular partial remission (nPR), or confirmed partial remission (PR) based on the 2008 Modified International Workshop on Chronic Lymphocytic Leukemia (IWCLL) National Cancer Institute-Working Group (NCI-WG) Guidelines criteria to the earliest date of progressive disease (PD) or death. DOR was analyzed by Kaplan-Meier (K-M) methodology.
Time Frame: as for outcome 25
Population: All enrolled participants who received at least one dose of venetoclax, had active disease at baseline, and achieved a response of PR or better
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 161
months | 36.0 [30.0 to 38.9]

28. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from the date of first dose of venetoclax to the date of earliest disease progression (PD). TTP was analyzed by Kaplan-Meier (K-M) methodology.
Time Frame: as for outcome 25
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
months | 43.0 [33.4 to 47.2]

29. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the number of days from the date of first dose of venetoclax to the date of earliest disease progression (PD) or death. PFS was analyzed by Kaplan-Meier methodology.
Time Frame: as for outcome 25
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
months | 35.5 [32.9 to 42.9]

30. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the number of days from the date of first dose of venetoclax to the date of death. For participants who did not die, their data was censored at the date of last study visit or the last known date to be alive, whichever was later. OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 25
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 210
months | NA [53.1 to NA] — Not calculable/estimable due to low number of participants with events

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was 184 weeks. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean duration on study drug was 123 weeks.
Arm/Group | Venetoclax
All-Cause Mortality (participants affected / at risk) | 65/210
Serious Adverse Events (participants affected / at risk) | 106/210
Other Adverse Events (participants affected / at risk) | 179/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax (N=210)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
EVANS SYNDROME (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 (7)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 (6)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
CATARACT CORTICAL (Eye disorders) | 1 (1)
CATARACT NUCLEAR (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 10 (15)
SUDDEN DEATH (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1 (1)
ACUTE SINUSITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 3 (5)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FUNGAL SEPSIS (Infections and infestations) | 1 (2)
HAEMOPHILUS INFECTION (Infections and infestations) | 2 (2)
HERPES VIRUS INFECTION (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1)
INFLUENZA (Infections and infestations) | 4 (4)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1)
LIVER ABSCESS (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
MENINGITIS ASEPTIC (Infections and infestations) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 21 (26)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 (1)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 2 (3)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 2 (2)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (2)
SALMONELLOSIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SERRATIA SEPSIS (Infections and infestations) | 1 (2)
STREPTOCOCCAL INFECTION (Infections and infestations) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
INJURY (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 (5)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OESOPHAGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SKIN SQUAMOUS CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
SQUAMOUS CELL CARCINOMA OF HEAD AND NECK (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
BRAIN OEDEMA (Nervous system disorders) | 1 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (2)
HEADACHE (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (2)
PRESYNCOPE (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (2)
RENAL COLIC (Renal and urinary disorders) | 1 (2)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 (1)
STEM CELL TRANSPLANT (Surgical and medical procedures) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax (N=210)
ANAEMIA (Blood and lymphatic system disorders) | 26 (33)
NEUTROPENIA (Blood and lymphatic system disorders) | 90 (189)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 39 (60)
CONSTIPATION (Gastrointestinal disorders) | 18 (19)
DIARRHOEA (Gastrointestinal disorders) | 66 (105)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 12 (13)
NAUSEA (Gastrointestinal disorders) | 35 (42)
VOMITING (Gastrointestinal disorders) | 15 (20)
FATIGUE (General disorders) | 15 (18)
OEDEMA PERIPHERAL (General disorders) | 11 (11)
PYREXIA (General disorders) | 19 (24)
BRONCHITIS (Infections and infestations) | 18 (24)
PNEUMONIA (Infections and infestations) | 11 (12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 58 (113)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 12 (12)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 13 (13)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 11 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 21 (22)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 (16)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (17)
HEADACHE (Nervous system disorders) | 18 (23)
INSOMNIA (Psychiatric disorders) | 13 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 (24)
RASH (Skin and subcutaneous tissue disorders) | 16 (18)
HYPERTENSION (Vascular disorders) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02980731/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02980731/SAP_001.pdf